CLINICAL TRIAL: NCT00283764
Title: A Phase 3, 12-Week, Parallel-Design Study Comparing The Safety, Efficacy, and Ease Of Use Of Xalatan When Self-Administered By Subjects With Open-Angle Glaucoma Or Ocular Hypertension Using Either A Conventional Dropper Bottle Or A Forced-Flow Delivery Device
Brief Title: Safety And Efficacy Of Xalatan Delivered Using Either A Conventional Dropper Bottle or A Delivery Device
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A6111086
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2015-03

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

INTERVENTIONS:
Drug: Xalatan

SUMMARY:
Compare the antihypertensive efficacy of two methods for instilling Xalatan eyedrops

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma or ocular hypertension in 1 or both eyes

Exclusion Criteria:

* History of closed/barely open anterior chamber angle or a history of angle closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure (IOP) level in the study eye.

SECONDARY OUTCOMES:
Successful eyedrop self-deliveries
Ease of eyedrop administration
Change in safety assessments throughout the study period
Subject preference for the method of drop delivery

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer